CLINICAL TRIAL: NCT05432765
Title: AIIM Trial: Protecting Kidney Function After Transplantation Using Augmented Intelligence Based Immunosuppression Dosing
Brief Title: AIIM Trial: Personalized Medicine Approach to Kidney Allograft Function
Acronym: AIIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202201106
Record Dates: First submitted 2022-06-06; First posted 2022-06-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Kidney Transplant Rejection
Keywords: Kidney; Transplant; dd-cf DNA; Personalized Medicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients who meet eligibility criteria will be randomized (1:1) into one of two treatment arms using balanced-permuted block randomization with a block size of 4, stratified by transplant number (first versus second). The random allocation sequence will be prepared by the study statistician and implemented automatically by the randomization procedure in REDCap
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physician Dosing (Active Comparator): Subjects will continue per SOC, where the management of their immunosuppression regimen will be determined by their physician per center practices, including dd-cfDNA data.
  Interventions: Other: Standard of Care Dosing
- PPM Dosing (Experimental): Subjects will have dd-cfDNA data analyzed by PPM. Data, such as drug levels and regimens, will be used to fit a 2nd order polynomial for each patient to build patient-specific dose-response profiles with covariates that include the administered drugs tacrolimus, steroids, and MMF/MPA. PPM will be used to derive an optimal combination of tacrolimus, MMF/MPA, and prednisone to achieve minimal renal allograft injury, while staying within the therapeutic range of the medications. All else being equal, the most efficacious combination with the lowest dose of tacrolimus will be utilized.
  Interventions: Other: Phenotypic Personalized Medicine Dosing

INTERVENTIONS:
Other: Phenotypic Personalized Medicine Dosing — Phenotypic Personalized Medicine (PPM) will mediate mechanism-independent and patient specific optimization of immunosuppression. We have developed a powerful platform that allows the provider to use clinical data to construct a Parabolic Response Surface (PRS). Using this visualization of the data, the provider can them make a decision on the optimal combination of drug doses needed to achieve the desired outcome.
  Arms: PPM Dosing
Other: Standard of Care Dosing — Providers will decide on the combination of drug doses needed based on their overall assessment per standard of care.
  Arms: Physician Dosing

SUMMARY:
The objective of the proposed study it to perform a pilot clinical trial both to establish feasibility of applying a computational, augmented intelligence based approach, Phenotypic Precision Medicine (PPM), to optimizing combination drug therapy and to gather preliminary data to support a larger fully powered multi-center clinical trial. The key rationale for this clinical selection is that we have the technical, biological, and medical expertise in this disease, a wealth of experience in the use of PPM in both in vitro and the clinical setting, and a robust and integrated transplant program with a well-functioning clinical trial infrastructure.

DETAILED DESCRIPTION:
In this pilot/feasibility trial the investigators will assess the feasibility of the trial design described below and perform a pilot study to obtain information for the design of a future multicenter randomized controlled trial (RCT). These goals will be achieved within the three year span of this program. The study has organized the investigator team to be able to achieve the following goals: 1) obtain regulatory approval, 2) optimize the clinical trial design, 3) recruit patients, 4) conduct the study, including optimization of immunosuppression regimen and monitoring the endpoints of interest, 5) conduct statistical analysis of the results, and 6) analyze the findings. Thirty-four subjects will be recruited at the time of kidney transplantation. Inclusion and exclusion criteria are listed below. All subjects will be started with institutional standard of care (SOC): quadruple immunosuppressive therapy with in-duction (basiliximab or antithymocyte globulin), tacrolimus, steroids, and mycophenolate mofetil/mycophenolic acid (MMF/MPA). Maintenance immunosuppression after transplantation will also be determined by the center per SOC. At recruitment, one month after transplantation, subjects without biopsy proven rejection will be recruited and enrolled in the baseline monitoring period of the study. Monitoring includes weekly dd-cfDNA (donor-derived cell-free DNA) measurements, drawn at the same time as SOC labs, up to three months after transplantation. Subjects will continue to be seen per clinical SOC Both SOC and dd-cfDNA labs will be obtained per patient preference (commercial lab, mobile phlebotomy, or at UF). Dd-cfDNA assessments will be performed at a Clinical Laboratory Improvement Amendments (CLIA)-approved centralized location per company standards. Clinical SOC includes an updated history and physical, including a full medication history, biochemical and hematological measurements, and drug exposure of tacrolimus monitored by obtaining trough level measurements. Three months after transplantation, a graft biopsy will be obtained and analyzed by an expert renal pathologist. Patients with evidence of rejection on biopsy will be excluded. Patients without rejection (Banff Classification 2018 active or chronic cellular or antibody mediated rejection) will undergo balanced randomization (1:1) to one of the following treatment arms:

1. Control arm: Subjects will continue per SOC, where the management of their immunosuppression regimen will be determined by their physician per center practices, including dd-cfDNA data.
2. Treatment arm: Subjects will have dd-cfDNA data analyzed by PPM. Data, such as drug levels and regimens, will be used to fit a 2nd order polynomial for each patient to build patient-specific dose-response pro-files with covariates that include the administered drugs tacrolimus, steroids, and MMF/MPA. PPM will be used to derive an optimal combination of tacrolimus, MMF/MPA, and prednisone to achieve minimal renal allograft injury, while staying within the therapeutic range of the medications. All else being equal, the most efficacious combination with the lowest dose of tacrolimus will be utilized.

In either arm, if a change is made in the immunosuppression regimen, SOC and dd-cfDNA labs will be obtained one week later to assess for changes and for the regimen to be adjusted accordingly. If no change is made in the immunosuppression regimen, the subject will continue with their SOC labs and clinic visit schedule. All subjects will undergo a protocol biopsy at the completion of the study at 15 months (12 months after first biopsy).

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older) patients with end-stage renal disease (ESRD)
* Recipient of a first or subsequent deceased donor kidney transplant
* Clinical indication to receive tacrolimus as the primary immunosuppression
* Willing and able to provide written informed consent to participate

Exclusion Criteria:

* Recipients of transplanted organs other than kidney
* Recipients of a transplant from a monozygotic (identical) sibling
* Human Leukocyte Antigen (HLA)-identical donor (zero out of six antigen mismatch donor)
* Recipient of third or more transplant
* Current or historical panel reactive antibodies of more than 50%
* Blood Type (ABO) incompatibility or known moderate or strong donor specific antibodies
* De novo or recurrent glomerulonephritis on 3-month biopsy
* Lupus nephritis on 3-month biopsy
* Focal segmental glomerulosclerosis on 3-month biopsy
* BK polyomavirus nephropathy in current or prior transplant
* Recipient of a bone marrow transplant
* Recipient who is pregnant
* Enrollment in a competing trial that would interfere with selection or alteration of immunosuppression
* Inability to follow up with transplant center for up to 15 months after transplantation
* Anticipated major surgery during the time of planned study
* Major medical illness with life expectancy less than 15 months
* Suspicion of noncompliance
* Anticipated relocation to a location that would not allow follow up at local center in the next 18 months
* Inability to tolerate normal range levels of tacrolimus

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2030-08-12 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in renal allograft interstitial fibrosis (IF) between 3-month baseline up to 15-month follow-up. | Change from 3-month baseline to 15-month follow-up
  Multiple studies have used this outcome because it 1) correlates well with renal function as measured by Creatinine Clearance (CrCl), 2) is a quantitative, continuous, and objective measure, thus needing fewer subjects to show a difference between groups in a small study, and 3) it is less susceptible to acute fluctuations than CrCl and more reflective of chronic injury. Renal allograft IF is a continuous variable that ranges from 0 to 100%.

SECONDARY OUTCOMES:
Change in Creatinine Clearance | Change from 3-month baseline to 15-month follow-up
  This is a quantitative measure of kidney function.
Change in tubular atrophy and vacuolization on biopsy | Change from 3-month baseline to 15-month follow-up
  Used as markers of allograft function and chronic allograft injury.
24-hour proteinuria | Change from 3-month baseline to 15-month follow-up
  This would be performed using a 24-hour urine collection method for the greatest accuracy.
Cumulative tacrolimus exposure | At 15-month follow-up
  Measured by a summation of total tacrolimus dose over the 12 months of study dosing and by the integration of the cumulative tacrolimus trough levels over the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zarrinpar, MD PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Shands, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will use methods in place from previous and ongoing studies to customize a data management system for the AIIM Trial. Data from study visits will be acquired on paper and processed using a REDCap database provided by the UF Clinical and Translational Science Institute and stored on secure UF servers. Initial examination of data will include descriptive statistics, frequency distributions, and histograms to identify outliers and missing data and to check data source adequacy. This process will be supervised by the PI and lead statistician. Any entry error and/or inconsistency will be discussed during meetings with the study team. Quarterly statistical summaries and progress reports will be generated by the statisticians for review by all investigators. This will be delivered in the form of a web-based platform using the R Shiny app to closely monitor participants accrual and maximize data quality.

REFERENCES:
- [Result] Zarrinpar A, Busuttil RW. Liver transplantation: past, present and future. Nat Rev Gastroenterol Hepatol. 2013 Jul;10(7):434-40. doi: 10.1038/nrgastro.2013.88. Epub 2013 Jun 11. PMID 23752825
- [Result] Starzl TE, Iwatsuki S, Shaw BW Jr, Gordon RD, Esquivel CO. Immunosuppression and other nonsurgical factors in the improved results of liver transplantation. Semin Liver Dis. 1985 Nov;5(4):334-43. doi: 10.1055/s-2008-1040630. PMID 3909427
- [Result] Tanzi MG, Undre N, Keirns J, Fitzsimmons WE, Brown M, First MR. Pharmacokinetics of prolonged-release tacrolimus and implications for use in solid organ transplant recipients. Clin Transplant. 2016 Aug;30(8):901-11. doi: 10.1111/ctr.12763. Epub 2016 Jun 18. PMID 27220013
- [Result] Marcen R. Immunosuppressive drugs in kidney transplantation: impact on patient survival, and incidence of cardiovascular disease, malignancy and infection. Drugs. 2009 Nov 12;69(16):2227-43. doi: 10.2165/11319260-000000000-00000. PMID 19852526
- [Result] Williams D, Haragsim L. Calcineurin nephrotoxicity. Adv Chronic Kidney Dis. 2006 Jan;13(1):47-55. doi: 10.1053/j.ackd.2005.11.001. PMID 16412970
- [Result] di Paolo S, Teutonico A, Stallone G, Infante B, Schena A, Grandaliano G, Battaglia M, Ditonno P, Schena PF. Cyclosporin exposure correlates with 1 year graft function and histological damage in renal transplanted patients. Nephrol Dial Transplant. 2004 Aug;19(8):2107-12. doi: 10.1093/ndt/gfh344. Epub 2004 Jun 8. PMID 15187199
- [Result] Fortin MC, Raymond MA, Madore F, Fugere JA, Paquet M, St-Louis G, Hebert MJ. Increased risk of thrombotic microangiopathy in patients receiving a cyclosporin-sirolimus combination. Am J Transplant. 2004 Jun;4(6):946-52. doi: 10.1111/j.1600-6143.2004.00428.x. PMID 15147429
- [Result] U.S. Multicenter FK506 Liver Study Group. A comparison of tacrolimus (FK 506) and cyclosporine for immunosuppression in liver transplantation. N Engl J Med. 1994 Oct 27;331(17):1110-5. doi: 10.1056/NEJM199410273311702. PMID 7523946
- [Result] Ekberg H, Grinyo J, Nashan B, Vanrenterghem Y, Vincenti F, Voulgari A, Truman M, Nasmyth-Miller C, Rashford M. Cyclosporine sparing with mycophenolate mofetil, daclizumab and corticosteroids in renal allograft recipients: the CAESAR Study. Am J Transplant. 2007 Mar;7(3):560-70. doi: 10.1111/j.1600-6143.2006.01645.x. Epub 2007 Jan 22. PMID 17229079
- [Result] Ekberg H, Bernasconi C, Tedesco-Silva H, Vitko S, Hugo C, Demirbas A, Acevedo RR, Grinyo J, Frei U, Vanrenterghem Y, Daloze P, Halloran P. Calcineurin inhibitor minimization in the Symphony study: observational results 3 years after transplantation. Am J Transplant. 2009 Aug;9(8):1876-85. doi: 10.1111/j.1600-6143.2009.02726.x. Epub 2009 Jun 26. PMID 19563339